CLINICAL TRIAL: NCT02744313
Title: MR Imaging of Fat Deposition in Adolescents With First Time Antipsychotic Use
Status: Completed | Type: Observational
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: American Academy of Child Adolescent Psychiatry. (Other)
Responsible Party: Principal Investigator, Margaret Hahn, MD, PhD, FRCPC, Centre for Addiction and Mental Health
Other Study IDs: 060/2014
Record Dates: First submitted 2016-04-06; First posted 2016-04-20 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Adiposity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Antipsychotic serum levels, GLP-1, glucagon, cytokines, c-peptide
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AP Naive: Group followed over 12 weeks to measure fat deposition, insulin resistance, and glucose tolerance.

SUMMARY:
This study will focus on a population of antipsychotic (AP) naïve adolescents and young adults and will measure fat accumulation in relation to exposure to atypical antipsychotic medications.

DETAILED DESCRIPTION:
Atypical Antipsychotics (AAPs) are known to cause metabolic dysfunction, and adolescents are especially vulnerable to this effect. The anthropometric measures routinely used to monitor these metabolic side effects may, in fact, underestimate risk in the pediatric population as they are not a good index of hepatic and visceral adipose tissue.

This study will measure fat accumulation over a 12 week period in adolescents and young adults taking an AAP for the first time. MRI imaging will measure hepatic, and visceral adipose tissue at baseline and study end. An Oral Glucose Tolerance Test will measure glucose resistance and insulin sensitivity. In an exploratory fashion, investigators will also image the brain to assess for volumetric changes which may occur in association with AAP treatment and changes in metabolic indices.

ELIGIBILITY:
Inclusion Criteria:

* AP naïve or AP-free for 3 months or greater
* prescribed an AP for treatment
* age 12-35
* using contraceptive (females of child bearing age)

Exclusion Criteria:

* currently taking AP or been taking AP for greater than 1 week within the past 3 months
* pregnant or planning to become pregnant
* eating disorder (active or previous)
* clinical or laboratory evidence of uncompensated cardiovascular, endocrine, haematological, or pulmonary disease
* major medical or surgical event in the preceding 3 months
* acute suicidal risk

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants recruited will be selected from clinical settings. Participants will be flagged by their care provider and offered the opportunity to participate should they meet criteria. As well, participants who are interested in the study and may meet criteria can refer themselves to the study.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2016-04; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change in hepatic and visceral adipose tissue from baseline to 3 months | Baseline and 3 months
  Adipose tissue is measured by an MRI. Fat content will be compared between baseline and study end (3 months).

SECONDARY OUTCOMES:
Change in glucose tolerance from baseline to 3 months. | Baseline and 3 months
  An Oral Glucose Tolerance Test (OGTT) will measure these outcomes at baseline and study end (3 months). Glucose is measured fasting (mmol/L) at the start of the OGTT and then 2 hours post glucose drink.
Change in insulin sensitivity from baseline to 3 months. | Baseline and 3 months
  An Oral Glucose Tolerance Test (OGTT) will measure these outcomes at baseline and study end (3 months). Insulin is measured fasting (pmol/L) at the start of the OGTT and then 2 hours post glucose drink.
Body Mass Index (BMI) | Baseline, 4 weeks, 8 weeks, 12 weeks
  BMI in kg/m^2
Change in appetite | Baseline and 3 months
  Visual analog scale
Change in weight | Baseline, 4 weeks, 8 weeks, 12 weeks
  Weight in kilograms

OTHER OUTCOMES:
Quality of life | Baseline and 3 months
  Assessed with the Pediatric Quality of Life (PedsQL) self-report questionnaire. Items are rated from 1 to 5, with a score of 5 indicating higher levels of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Hahn, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre For Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world — http://www.camh.ca/en/research